CLINICAL TRIAL: NCT00413985
Title: Growth and Development in Preterm Infants Fed Human Milk Containing a Powdered Human Milk Fortifier (HMF) Post Hospital Discharge
Brief Title: Post Discharge Human Milk Fortifier in Preterm Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Deborah O'Connor, Associate Chief, Clinical Dietetics, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1000003971
Record Dates: First submitted 2006-12-19; First posted 2006-12-20 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Infant, Low Birth Weight
Keywords: Low Birth Weight; Fortified Human Milk; breastfeeding; infants; growth
MeSH Terms: conditions — Breast Feeding

INTERVENTIONS:
Drug: Nutrient-enriched human milk

SUMMARY:
The purpose of this study is to determine whether low birth weight (LBW) infants fed human milk (HM)supplemented with a specially designed powdered human milk fortifier until 12 weeks after hospital discharge will have better growth and neurodevelopment than infants fed HM alone.

DETAILED DESCRIPTION:
Consensus exists in the literature that a significant proportion of low birth weight (LBW, <1800 g) infants leave hospital with overt signs of under-nutrition (eg. growth retardation). Recent evidence from randomized control trials suggest that provision of nutrient-enriched feeding to formula-fed premature infants after hospital discharge improves their growth, accretion of lean body mass and bone mineral content compared to infants fed a standard term formula. While available data suggest an advantage of human milk feeding after hospital discharge, experimental evidence on which to base guidelines to enrich, or not to enrich, human milk (HM) are notably absent.

ELIGIBILITY:
Inclusion Criteria:

* Birth Weight between 750-1800 g
* Gestational Age at birth between 26 and 32 weeks
* Singleton or twin birth (for twins to be eligible, both must meet eligibility criteria)
* Small for Gestational age or appropriate for gestational age
* ≥ 80% energy received from human milk in the previous three days
* ≥ 25% of human milk consumed orally in the previous three days
* Mother agrees to exclusively feed her infant human nilk after discharge
* If so randomized, parents agree to supplement ~1/2 or the human milk provided to her infant as powdered human milk fortifier for 12 weeks after hospital discharge
* Subject's parents have voluntarily signed an informed consent form

Exclusion Criteria:

* Serious congenital or chromosomal anomalies that will affect growth
* Grade III or IV periventricular/intraventricular hemorrhage
* Received steroids within 14 days o randomization
* Asphyxia (hypoxia or ischemia) es evident by severe and permanent neurological data
* Maternal incapacity, including maternal cocaine or alcohol abuse dring pregnancy, or concurrent, or mother or infant has tested positive for HIV
* Principal residence of study family outside GTA
* Mother unable to verbally communicate in English
* A single feeding must be fortified > 24 kcal/oz or >50% of feeds need to be fortified

Ages: 1 Day to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40
Dates: Start 2004-01; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Growth (weight, length and head circumference)
Body composition (fat-free mass, whole body mineral content, fat mass
Milk consumption
Estimated energy and nutrient intakes
Duration/exclusivity of breastfeeding
Morbidity (serious adverse events, hospital re-admissions)
Development (mental, motor, visual and language)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah L O'Connor, RD, PhD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (9):
- Canada (9):
  - The Credit Valley Hospital, Mississauga, Ontario
  - Rouge Valley Centenary, Toronto, Ontario
  - The Scarborough Hospital, Toronto, Ontario
  - Toronto East General Hospital, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Sunnybrook and Women's Health Sciences Centre, Toronto, Ontario
  - St. Joseph's Health Centre, Toronto, Ontario

REFERENCES:
- [Derived] O'Connor DL, Khan S, Weishuhn K, Vaughan J, Jefferies A, Campbell DM, Asztalos E, Feldman M, Rovet J, Westall C, Whyte H; Postdischarge Feeding Study Group. Growth and nutrient intakes of human milk-fed preterm infants provided with extra energy and nutrients after hospital discharge. Pediatrics. 2008 Apr;121(4):766-76. doi: 10.1542/peds.2007-0054. PMID 18381542